CLINICAL TRIAL: NCT04200027
Title: Robotic vs. TaTME Rectal Surgery (ROTA STUDY) Matched Cohort Trial for Mid to Low Rectal Cancer Surgery Evaluation Trial in the Hands of an Experienced Surgeon
Brief Title: Robotic vs. TaTME Rectal Surgery (ROTA STUDY)
Acronym: ROTA
Status: Not yet recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Issam al-Najami, principal investigator. phd. associate professor, Odense University Hospital
Other Study IDs: svb IAN 151119
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robotic total mesorectal Excision: robotic assissted total mesorectal excision
  Interventions: Procedure: total mesorectal excision
- Transanal total mesorectal excision: Transanally assissted total mesorectal excision
  Interventions: Procedure: total mesorectal excision

INTERVENTIONS:
Procedure: total mesorectal excision — Total Mesorectal Excision Total Mesorectal Excision is currently the standard technique for surgical treatment of RC. It was first described in 1982 by Bill Heald, and relies on the excision of the whole mesorectum within an intact mesorectal fascia, with the contained lymphatic system along with the tumour bearing bowel segment Total mesorectal excision

SUMMARY:
Background Recent novel surgical techniques for resection of low rectal cancer have been introduced and these approaches have the potential to overcome anatomical limitations like obesity, narrow male pelvis and bulky and low tumours. Two of these procedures are robotic low anterior resection (RLAR) and transanal total mesorectal excision (TaTME).

Both approaches have distinct advantages and limitations however there have been no head to head trial comparing RLAR and TaTME for patients with mid to low rectal cancer undergoing surgery by experienced surgeons. Previous studies looking at the oncological outcomes of either TaTME or robotic TME included many centres where the surgeons were on a learning curve and hence the true oncological outcomes and clinical benefits cannot be measured accurately.

The primary objective of this pilot study is to conduct a multicentre prospective trial to investigate clinical outcomes, in particular disease free survival (DFS) in patients undergoing RLAR and TaTME. The additional goal is to investigate other efficacy measures, complications rates, recruitment feasibility and protocol refinement.

Method

This pilot study will be a prospective, observational, case-matched, two -cohort, multicentre designed to investigate the oncological and clinical outcomes of patients with mid-to-low, non-metastatic rectal cancer undergoing low anterior resection (LAR) using robot-assisted surgery ( RLAR), or transanal total mesorectal excision (TaTME).

The inclusion criteria consist of experienced surgeons defined as 60 prior procedures with RLAR or TaTME to meet the enrolment criteria for the RLAR and TaTME arm, respectively. Successful oncological and clinical outcomes are defined as circumferential resection margin (CRM) ≥1 mm with minimal postoperative morbidity (absence of Clavien-Dindo grade III-IV complications within 30 days after surgery). Local and distal recurrence rates with DFS over 3 years will be measured as primary outcome.

Secondary and exploratory endpoints will include length of hospital stay, intraoperative time, intraoperative blood loss, harvested lymph nodes, distal resection margin, incompleteness of mesorectum, CRM involvement, unplanned conversion rates, 30-days postoperative complications and overall recurrence rate. The Quality of life assessment questionnaires will be performed preoperatively, 6 months and 12 months after reversal of ileostomy.

Propensity score matching will be used to minimize bias from the nonrandomized treatment assignment. The RLAR and TaTME cohorts will be matched by propensity scores accounting for factors significantly associated with either undergoing robotic surgery or TaTME occurrence on logistic regression analysis.

Ethics and Dissemination The medical ethical committees of all the participating countries will be involved in approving the study protocol. Results of the primary and secondary end points will be submitted for publication in peer-reviewed journals.

DETAILED DESCRIPTION:
Introduction Colorectal cancer (CRC) is the fourth most common malignant disease with over 1 million new cases each year worldwide (1) The outcome of surgery for rectal cancer has improved substantially during the past two decades due to TME, which involves complete removal of the mesorectum with preservation of the pelvic autonomic nerves. Local recurrence rate of rectal cancer has fallen sharply because radially spread cancer cells in the mesorectum are removed by complete resection of this tissue.(2)(3)(4) Minimally invasive surgery (MIS) is slowly taking over as the preferred operative approach for colorectal diseases. Recently published randomized clinical trials (RCTs), such as COLOR II, COREAN and CLASICC, have shown better results for laparoscopic total mesorectal excision (in terms of short-term and long-term outcomes), when compared with open TME(5)(6)(7) However the utility of laparoscopic TME is limited in patients with low rectal cancer, who require surgeons with experience in ultra-low sphincter-saving laparoscopic surgery, which has a high risk of leaving a positive circumferential resection margin (CRM). In addition, narrow pelvic anatomy; male sex and high body mass index (BMI) are also unfavourable patient characteristics for a laparoscopic approach

The need to overcome these challenges has motivated surgeons to adopt alternative techniques. The two more recent procedures that have been introduced to surgical management of rectal cancer are robotic low anterior resection (RLAR) and Transanal Total Mesorectal Excision (TaTME). These two new procedures have the potential to overcome anatomical limitations like obesity, narrow male pelvis and bulky and low tumours to improve surgical treatment and thereby potentially oncological outcomes.

TaTME combines the TAMIS ( transanal minimally invasive surgery ) and trans-abdominal approaches in order to achieve TME.Transanal TME (TaTME) typically starts with the rectal resection and progresses to the splenic flexure/sigmoid colon mobilization in a "bottom-up" manner (8). A single-incision laparoscopic surgery port is introduced into the anal canal to gain endoscopic access to the rectum, pneumorectum is established, A purse-string suture is applied below the tumor, and this ensures an adequate oncological distal margin (9). Transanal excision is subsequently performed using laparoscopic instruments Rectal distension with CO2 combined with magnified optics permits excellent visualization of tissue planes. Easier access to the low rectum aid the surgeon with better quality TME and precise selection of the distal resection margin under direct visualization helps ensure an adequate margin. TaTME may potentially aid to a safer anastomosis by avoiding the multiple stapler firings often required in the laparoscopic approach and may result in higher rates of sphincter preserving surgery.

Robotic approach has been subject to much interest in recent years from its potential learning benefits to the operating surgeon and clinical benefits to the patients. Some of the clinical benefits include shorter hospital stay and improved functional outcomes compared to laparoscopic surgery (10) The other advantages provided by the robotic platform hold the potential to provide improved clinical outcomes, (11)(12) (13).

Both of the new procedures have been compared retrospectively to open and conventional laparoscopic surgery in various trials, which show that these methods are safe and feasible (9)(14). However, data on direct comparison of these two techniques are still lacking.

Potential benefits of robotic rectal resections Technical Benefits The potential benefits of robotic systems over laparoscopic TME include superior three-dimensional vision, seven degrees of freedom of movement replicating the surgeon's hand movements, lack of tremor and potential superior ergonomics, suggesting potential application in both routine and more difficult cases

Operator Learning Benefits The main criticisms of robotic TME are the longer operating times and notable trends of higher costs, compared to laparoscopic TME(14). Greater use of and familiarity with the robotic system has led to significant improvements operation time, rates of conversion to open surgery and the number of harvested lymph nodes.

Bokhari et al (15) suggested that the learning curve of robotic colorectal surgery was achieved at 15 to 25 cases with 3 learning phases after analysing 50 patients by using cumulative sum (CUSUM ) method. The author suggested that Phase 3 was achieved after 25 cases and this represented a mastery phase in which more challenging cases can be managed. Kim et al showed that the learning curve plateaued after 65 cases for early Laparoscopic TME as opposed to after 32 cases for Robotic TME (16) Most studies to date about RLAR were done using the da Vinci Si system or older models. With the newer systems X or Xi, and once the surgeons have achieved at least 60 procedures we believe that the outcomes and operating time is less, that has been recently published by the ROLAR trial (12). Similarly to achieve good clinical and oncological outcomes with TaTME surgeons are required to have performed at least 60 cases. Hence we decided to choose 60 procedures as an arbitrary number to select our surgeons experience involved in this trial. Selecting this number suggest that the surgeons are in a mastery period and hence are expected to have good clinical and oncological outcomes Considering the paucity of evidence on direct comparison of these two procedures we aim to directly compare both procedures for the disease free survival and other clinical and oncological outcomes in the hands of experienced surgeons.

Potential benefits of TaTME rectal resections TaTME offers better access to the lower rectum even in a difficult pelvis and also ensure a clear distal margin with insertion of a distal to the tumour purse string under direct vision. This ensures an end-to-end anastomosis without the need of multiple stapler firings. This approach also allows two-team synergy with an abdominal and perineal surgeon operating simultaneously.

The technique however still requires significant surgical skills and the abilty to operate in a confined space and concerns have been expressed about the spillage of tumour cells with direct handling and instrumentation.

Methods and analysis Design This is an observational prospective, multicentre trial. Patients will be assigned either RLAR or TaTME depends on the chosen centres.The centres would be doing either TaTME or RLAR for rectal cancer management. The study will include 330 patients from UK and Denmark. This study has no impact on staging investigations, timing of surgery or any other aspect of the patients' pre, peri or post-operative care. All decisions remain with the local clinician multi-disciplinary team including when to discharge from hospital. However, the biostatisticians performing the analysis will be blinded to the intervention

Objectives Outcome Measures Time point(s) of evaluation of this outcome measure (if applicable) Primary Objective The primary aim of the study is to compare the 3 year disease free survival between RLAR and TaTME in the hands of an experienced surgeon 3 year disease free survival 6 monthly post op for the first 2 years and 12 -monthly follow-up for next 3 years Secondary/ exploratory Objectives Surgical morbidity/mortality up to 90 days

Pathological quality assessment

Assessment of intraoperative adverse events within advanced minimally-invasive surgery

Overall survival at 3 years

Health economics assessments

Evaluation of the operative length of time

Recruitment per month per centre for the RLAR and TaTME ARMS

Completeness of mesorectum excision (TME) will be assessed by the pathologist and is defined as:

1. Distal resected margin ≥ 1cm
2. Lymph node yield
3. Mesorectalplane of surgery
4. R0 resection (all margins clear) To report "near misses" and associated impact upon clinical outcomes

Healthcare resource utilization (costs) including hospital length of stay, ICU hours, and productivity losses collected through a Labour Force survey). Return to work/activity will also be included Total OR utilisation time and operative time skin to skin, minutes This will be used as part of the feasibility assessment to determine the duration of the recruitment period and the follow-up phase. Patients dropout rate during follow-up will also be monitored Study population Participants with rectal cancer who are scheduled for initial treatment by TME.The inclusion and exclusion criteria are shown in Table 1 Table 1 Inclusion criteria Exclusion criteria

* Participant is willing and able to give informed consent for participation in the trial.
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* Male or Female, aged 18 years or above.
* Participant with life expectancy of less than 6 months.
* Undergoing TME surgery for rectal cancer after MDT discussion.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participant has no contra-indication to pelvic radiotherapy at the time of enrolment.
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Tumour distance from anal verge - 12 cm or less
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.

The Number of Participants The primary study end point, DFS is defined as the time following successful surgery to the first date of local, regional/distant relapse or death due to colorectal cancer (patients with secondary malignancy will be censored). Overall survival is defined as the time following successful surgery to death.

In the TaTME, it is assumed that the DFS is 92% and in the RLAR arm 95% at 3 years. A non-inferiority margin of 90% is selected. Based on this estimation, sample size calculation has been done with a one-sided level of significance of 20% and a power of 80%. A total number of 330 patients is needed, 165 patients in the RLAR arm and 165 patients in the TaTME are required with a 10% loss to follow-up assumed.

DFS will be analysed on an intent-to-treat (per protocol) basis using a log-rank test after propensity matching analysis has been conducted; a secondary analysis of DFS will also performed be using a Cox proportional hazards regression model with the unmatched cohort (without adjustment of baseline characteristics, i.e. propensity score match) that allowed for the effect of treatment and include lists of covariate with a statistical interaction of alpha level of 20%.

Data Management Case report forms (CRFs) will be entered in a secured online page. Only authorized staff at sites will have access via an individual secure login username and password to enter the data. All paper CRFs must be completed, signed/dated and returned to the investigator. Data reported on each CRF should be consistent with the source data or discrepancies should be explained. If information is not known, this must be clearly indicated on the CRF. All missing or ambiguous data will be queried. All sections are to be completed.

All trial records will be archived and securely retained for at least 25 years.

Ethics and dissemination The trial will be performed in accordance with the recommendations guiding physicians in biomedical research involving human subjects, adopted by the 18th World Medical Association General Assembly, Helsinki, Finland and stated in the respective participating countries laws governing human research, and Good clinical Practice. The medical ethical committees of all participating countries will have to approve the study protocol prior to enrolling patients.

Discussion

To date studies on TaTME and robotic TME have focused mainly on short term outcomes and oncological endpoints such as specimen quality, circumferential resection margin involvement and the free distal margin(14,17,18) In a recent study comparing TaTME and Robotic TME, there were no differences in the incidence of poor quality resection including incomplete quality of TME and positive circumferential resection margin (CRM) in both groups. However the authors noted that distal resection margin (DRM) involvement was higher in the TaTME group.(17) They attributed this to the learning curve effect of TaTME. As discussed earlier, previous reports have noted that the learning curve for robotic TME was less than laparoscopic surgery, which in effect TaTME is still a laparoscopic "bottom up "approach.

Nonetheless, the long term oncological parameters for both procedures , including overall survival, disease-free survival and local recurrence, are yet to be clarified. Secondly, there have been significant concerns in regards to an increased recurrence rate after TaTME (19).The Norwegian group have noted an unexpected increase in local recurrence after TaTME of 9.5 % after a median of 11months after surgery(19).The reasons for their observations were unclear , despite that fact that their surgeons performing TaTME were experienced and were proctored and trained in England and Spain for the procedure.

In 1980 Knight and Griffen (20)publised their stapling technique for low rectal cancer anastomosis using linear and circular stapler.This has lead to the introduction of the double stapling technique(21). The advantage is that the distal segment of the bowel is not opened and this avoids spillage from the rectal stump.

The possibility of increased local recurrences in TaTME may be related to the rectal transection and air flow during dissection from the perineum. The rectal purse-string suture is never completely air tight and this will invariably lead to shredding of microscopic cancer cells in the pelvis and hence this may lead to an increase rate of local recurrence.During a robotic TME and the use of the articulating robotic stapler ,the rectal transection is precise and there are no leakage of microscopic cancer cells in the pelvis.

With these current issues in mind, we aim to compare the 3 year disease free survival and local recurrence rate of the two procedures performed by experienced surgeons who are beyond their learning curve . Only surgeons who have peformed more than 60 procedures in either TaTME or robotic TME will be selected .

ROTA study will be the first multicentre prospective trial comparing RLAR and TaTME in regards to disease free survival (DFS) and other clinical trials Applications for funding, ethics approval and protocol amendments will be required.

Conclusions There is an urgent need to assess the long oncological outcomes of newer surgical techniques for TME (TaTME & RLAR) This will allow recommendations to be made for tailor made treatment of RC.

ELIGIBILITY:
Inclusion Criteria:

* • Participant is willing and able to give informed consent for participation in the trial.

  * Male or Female, aged 18 years or above.
  * Undergoing TME surgery for rectal cancer after MDT discussion.
  * Participant has no contra-indication to pelvic radiotherapy at the time of enrolment.
  * In the Investigator's opinion, is able and willing to comply with all trial requirements.
  * Tumour distance from anal verge - 12 cm or less
  * Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.

Exclusion Criteria:

* • Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.

  * Participant with life expectancy of less than 6 months.
  * Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The primary study end point, DFS is defined as the time following successful surgery to the first date of local, regional/distant relapse or death due to colorectal cancer (patients with secondary malignancy will be censored). Overall survival is defined as the time following successful surgery to death.
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2021-11-15 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
oncological outcomes RLAR vs TaTMe | 3 year disease free survival
  The primary aim of the study is to compare the 3 year disease free survival between RLAR and TaTME in the hands of an experienced surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Issam al najami, phd, Principal Investigator — The Department of clinical research, University of Southern Denmark, Denmark
Locations (2):
- Issam al-Najami, Svendborg, Southern Denmark, Denmark
- Jim Khan, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
see detailed study description
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: november 2019-november 2022

REFERENCES:
- [Background] Wiseman M. The second World Cancer Research Fund/American Institute for Cancer Research expert report. Food, nutrition, physical activity, and the prevention of cancer: a global perspective. Proc Nutr Soc. 2008 Aug;67(3):253-6. doi: 10.1017/S002966510800712X. Epub 2008 May 1. PMID 18452640
- [Background] Heald RJ, Husband EM, Ryall RD. The mesorectum in rectal cancer surgery--the clue to pelvic recurrence? Br J Surg. 1982 Oct;69(10):613-6. doi: 10.1002/bjs.1800691019. PMID 6751457
- [Background] Heald RJ, Ryall RD. Recurrence and survival after total mesorectal excision for rectal cancer. Lancet. 1986 Jun 28;1(8496):1479-82. doi: 10.1016/s0140-6736(86)91510-2. PMID 2425199
- [Background] van der Pas MH, Haglind E, Cuesta MA, Furst A, Lacy AM, Hop WC, Bonjer HJ; COlorectal cancer Laparoscopic or Open Resection II (COLOR II) Study Group. Laparoscopic versus open surgery for rectal cancer (COLOR II): short-term outcomes of a randomised, phase 3 trial. Lancet Oncol. 2013 Mar;14(3):210-8. doi: 10.1016/S1470-2045(13)70016-0. Epub 2013 Feb 6. PMID 23395398
- [Background] Bonjer HJ, Deijen CL, Abis GA, Cuesta MA, van der Pas MH, de Lange-de Klerk ES, Lacy AM, Bemelman WA, Andersson J, Angenete E, Rosenberg J, Fuerst A, Haglind E; COLOR II Study Group. A randomized trial of laparoscopic versus open surgery for rectal cancer. N Engl J Med. 2015 Apr 2;372(14):1324-32. doi: 10.1056/NEJMoa1414882. PMID 25830422
- [Background] Jeong SY, Park JW, Nam BH, Kim S, Kang SB, Lim SB, Choi HS, Kim DW, Chang HJ, Kim DY, Jung KH, Kim TY, Kang GH, Chie EK, Kim SY, Sohn DK, Kim DH, Kim JS, Lee HS, Kim JH, Oh JH. Open versus laparoscopic surgery for mid-rectal or low-rectal cancer after neoadjuvant chemoradiotherapy (COREAN trial): survival outcomes of an open-label, non-inferiority, randomised controlled trial. Lancet Oncol. 2014 Jun;15(7):767-74. doi: 10.1016/S1470-2045(14)70205-0. Epub 2014 May 15. PMID 24837215
- [Background] Kang SB, Park JW, Jeong SY, Nam BH, Choi HS, Kim DW, Lim SB, Lee TG, Kim DY, Kim JS, Chang HJ, Lee HS, Kim SY, Jung KH, Hong YS, Kim JH, Sohn DK, Kim DH, Oh JH. Open versus laparoscopic surgery for mid or low rectal cancer after neoadjuvant chemoradiotherapy (COREAN trial): short-term outcomes of an open-label randomised controlled trial. Lancet Oncol. 2010 Jul;11(7):637-45. doi: 10.1016/S1470-2045(10)70131-5. Epub 2010 Jun 16. PMID 20610322
- [Background] Hompes R, Guy R, Jones O, Lindsey I, Mortensen N, Cunningham C. Transanal total mesorectal excision with a side-to-end stapled anastomosis - a video vignette. Colorectal Dis. 2014 Jul;16(7):567. doi: 10.1111/codi.12660. No abstract available. PMID 24801986
- [Background] Sun Y, Xu H, Li Z, Han J, Song W, Wang J, Xu Z. Robotic versus laparoscopic low anterior resection for rectal cancer: a meta-analysis. World J Surg Oncol. 2016 Mar 1;14:61. doi: 10.1186/s12957-016-0816-6. PMID 26928124
- [Background] Lee SH, Lim S, Kim JH, Lee KY. Robotic versus conventional laparoscopic surgery for rectal cancer: systematic review and meta-analysis. Ann Surg Treat Res. 2015 Oct;89(4):190-201. doi: 10.4174/astr.2015.89.4.190. Epub 2015 Sep 25. PMID 26448918
- [Background] Trastulli S, Farinella E, Cirocchi R, Cavaliere D, Avenia N, Sciannameo F, Gulla N, Noya G, Boselli C. Robotic resection compared with laparoscopic rectal resection for cancer: systematic review and meta-analysis of short-term outcome. Colorectal Dis. 2012 Apr;14(4):e134-56. doi: 10.1111/j.1463-1318.2011.02907.x. PMID 22151033
- [Background] Jayne D, Pigazzi A, Marshall H, Croft J, Corrigan N, Copeland J, Quirke P, West N, Rautio T, Thomassen N, Tilney H, Gudgeon M, Bianchi PP, Edlin R, Hulme C, Brown J. Effect of Robotic-Assisted vs Conventional Laparoscopic Surgery on Risk of Conversion to Open Laparotomy Among Patients Undergoing Resection for Rectal Cancer: The ROLARR Randomized Clinical Trial. JAMA. 2017 Oct 24;318(16):1569-1580. doi: 10.1001/jama.2017.7219. PMID 29067426
- [Background] Yang Y, Wang F, Zhang P, Shi C, Zou Y, Qin H, Ma Y. Robot-assisted versus conventional laparoscopic surgery for colorectal disease, focusing on rectal cancer: a meta-analysis. Ann Surg Oncol. 2012 Nov;19(12):3727-36. doi: 10.1245/s10434-012-2429-9. Epub 2012 Jul 3. PMID 22752371
- [Background] Penna M, Hompes R, Arnold S, Wynn G, Austin R, Warusavitarne J, Moran B, Hanna GB, Mortensen NJ, Tekkis PP; TaTME Registry Collaborative. Transanal Total Mesorectal Excision: International Registry Results of the First 720 Cases. Ann Surg. 2017 Jul;266(1):111-117. doi: 10.1097/SLA.0000000000001948. PMID 27735827
- [Background] Perez D, Melling N, Biebl M, Reeh M, Baukloh JK, Miro J, Polonski A, Izbicki JR, Knoll B, Pratschke J, Aigner F. Robotic low anterior resection versus transanal total mesorectal excision in rectal cancer: A comparison of 115 cases. Eur J Surg Oncol. 2018 Feb;44(2):237-242. doi: 10.1016/j.ejso.2017.11.011. Epub 2017 Nov 26. PMID 29249592
- [Background] Kwak JM, Kim SH. Current status of robotic colorectal surgery. J Robot Surg. 2011 Mar;5(1):65-72. doi: 10.1007/s11701-010-0217-8. Epub 2010 Oct 2. PMID 27637262
- [Background] Lee L, de Lacy B, Gomez Ruiz M, Liberman AS, Albert MR, Monson JRT, Lacy A, Kim SH, Atallah SB. A Multicenter Matched Comparison of Transanal and Robotic Total Mesorectal Excision for Mid and Low-rectal Adenocarcinoma. Ann Surg. 2019 Dec;270(6):1110-1116. doi: 10.1097/SLA.0000000000002862. PMID 29916871
- [Background] Penna M, Hompes R, Arnold S, Wynn G, Austin R, Warusavitarne J, Moran B, Hanna GB, Mortensen NJ, Tekkis PP; International TaTME Registry Collaborative. Incidence and Risk Factors for Anastomotic Failure in 1594 Patients Treated by Transanal Total Mesorectal Excision: Results From the International TaTME Registry. Ann Surg. 2019 Apr;269(4):700-711. doi: 10.1097/SLA.0000000000002653. PMID 29315090
- [Background] Larsen SG, Pfeffer F, Korner H. Author response to: Comments on: Norwegian moratorium on transanal total mesorectal excision. Br J Surg. 2019 Dec;106(13):1855. doi: 10.1002/bjs.11374. No abstract available. PMID 31747073
- [Background] Knight CD, Griffen FD. An improved technique for low anterior resection of the rectum using the EEA stapler. Surgery. 1980 Nov;88(5):710-4. PMID 7434211
- [Background] Cohen Z, Myers E, Langer B, Taylor B, Railton RH, Jamieson C. Double stapling technique for low anterior resection. Dis Colon Rectum. 1983 Apr;26(4):231-5. doi: 10.1007/BF02562484. PMID 6839891
- [Derived] Jootun R, Cuk P, Ellebaek M, Andersen PV, Salomon S, Baatrup G, Al-Najami I, Khan J. Robotic vs. TaTME Rectal Surgery (ROTA STUDY) Matched Cohort Trial for Mid to Low Rectal Cancer Surgery Evaluation Trial in the Hands of an Experienced Surgeon. Int J Surg Protoc. 2022 Feb 18;26(1):7-13. doi: 10.29337/ijsp.163. eCollection 2022. PMID 35280494